CLINICAL TRIAL: NCT04828551
Title: Noninvasive Biomarkers of Metabolic Liver Disease 1.1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of California, San Diego (Other); Foundation for the National Institutes of Health (Other)
Responsible Party: Principal Investigator, Anthony Samir, Radiologist, Service Chief, Body Ultrasound Imaging Services, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019P002092
Record Dates: First submitted 2021-03-24; First posted 2021-04-02 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Blood Specimen Collection; Medication Review

STUDY DESIGN:
Masking Description: Study participants will not be randomized to individual treatment groups. To ensure a uniform distribution of scanner combinations, participants will follow a block-allocation pattern with different scanner combinations for different participants, however, patients and operators will not be blinded to ultrasound scanners being used.
  All efforts will be made to keep ultrasound operators blinded to clinical and laboratory data, however, it is not believed that this will significantly affect the ultrasound acquisition. The Visit 2 operator will be asked to not review the Visit 1 exam results.
  Central analysts will be blinded to key clinical and laboratory findings to minimize potential bias. Blinding of the central analysts will be outlined in a separate Image Review Charter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MGH and UCSD Study subjects (Other): This study will enroll patients with suspected or confirmed diagnosis of NAFLD. Based on protocol-specified FIB-4 values, about one-third are expected to have low, one-third to have intermediate, and one-third to have high likelihood of advanced fibrosis.
  Sex: 50:50 - Note- no stratification will be done based on sex Age: ≥ 18 yrs Demographic group: Patients with a high probability of NAFLD based on the eligibility criteria General health status: Patients with suspected or confirmed diagnosis of NAFLD Geographic location: Boston, MA (greater metropolitan areas) and San Diego, CA (greater metropolitan areas)
  Interventions: Device: Ultrasound based shear wave speed and fat quantification methods; Diagnostic Test: Blood collection; Other: Physical measurements; Other: Clinical history and medication reviews

INTERVENTIONS:
Device: Ultrasound based shear wave speed and fat quantification methods — Ultrasound based imaging parameters will be collected from all patients in two visits. These will include but may not be limited to SWE results, Quantitative ultrasound parameters,where available,including Attenuation Coefficient, Backscatter Coefficient, Shear Wave Dispersion, Speed of Sound, Ultrasound derived fat fraction Conventional Bmode (gray-scale) and Doppler ultrasound images,including An image of the liver and right kidney on the same image for hepatorenal index calculation Right liver lobe for skin to liver capsule distance calculation Portal vein Doppler for portal vein pulsatility index measurement VCTE and Controlled Attenuation Parameter measurements with the Fibroscan system
Diagnostic Test: Blood collection — Blood will be collected by trained phlebotomists at each site using routine methods and standard collection tubes.
  Total volume is expected to be about 10 mL or less Blood collected at MGH will be analyzed by the MGH clinical laboratory. Blood collected at UCSD will be analyzed by the UCSD clinical laboratory. Blood results obtained within the 3-month interval prior to the screening visit at the MGH or UCSD laboratories will be considered acceptable for study analyses and may be used at PI discretion. For each laboratory, the normal ranges for each blood test will be recorded and filed
Other: Physical measurements — Height will be recorded at Screening. Weight and vital signs will be recorded at each visit. Body mass index will be calculated at each visit. All measurements will be made by trained coordinators using standard and calibrated instruments.
Other: Clinical history and medication reviews — The following questionnaires will be administered at Screening:
  Medical history questionnaire Medication use questionnaire Alcohol consumption questionnaire Physical activity questionnaire
  The following questionnaires will be administered at Visit 1 and Visit 2:
  Interim medical history questionnaire Change in medication use questionnaire Change in alcohol consumption will be recorded using a modified version of the alcohol use followback. Alcohol use for the 7 day period prior to Visit 1 and for all days between Visit 1 and Visit 2 will be recorded. Change in physical activity questionnaire

SUMMARY:
NIMBLE is a comprehensive collaborative effort to standardize, compare, validate, and advance the regulatory qualification of imaging and circulating biomarkers to diagnose and stage nonalcoholic steatohepatitis (NASH), and to predict and assess response to therapeutic intervention (https://fnih.org/what-we-do/biomarkers-consortium/programs/nimble). This study focuses on estimating the repeatability and reproducibility of ultrasound elastography-based biomarkers across a range of fibrosis stages.

DETAILED DESCRIPTION:
Study 1.1, is a prospective, two-center, short-term cross-sectional study to assess the reproducibility and repeatability of a set of specified ultrasound-based quantitative imaging biomarkers. The primary focus will be on imaging biomarkers of the liver fibrosis component of nonalcoholic fatty liver disease (NAFLD), rather than the steatosis or inflammation component. The rationale is that the fibrosis component is linked most closely to survival and other clinical outcomes. Study 1.1 will also collect data to explore vendor- or device-specific investigational biomarkers on other components of NAFLD such as steatosis and possibly inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years)
* Known or suspected NAFLD based on prior biopsy ≤ 36 months consistent with NAFLD OR
* Abnormal ALT (>30 U/L for men, > 19 U/L for women) without other common causes such as HCV, HBV, AND meets criteria within 36 months for ATP III criteria (2005 revision) for metabolic syndrome with any 3 of the 5:

Waist circumference (WC) > 102 cm (M) or > 88 cm (F)

* Fasting glucose ≥ 100 mg/dL or Rx
* TG≥150mg/dLorRx
* SBP > 130 mmHg
* DBP>85mmHg or Rx
* Able and willing to participate, including maintaining steady-state: physical activity, alcohol use, medications
* Classifiable into one of the following enrollment categories by FIB-4 (ALT, AST, platelets, date of birth) collected at screening visit if not available already within 3 months prior:

Low likelihood of advanced fibrosis: FIB-4 ≤ 1.3 (about one-third of enrolled participants, minimum 8, maximum 18), Intermediate likelihood of advanced fibrosis: 1.3 < FIB-4 < 2.67 (about one-third of enrolled participants, minimum 8, maximum 18), High likelihood of advanced fibrosis: FIB-4 ≥ 2.67: (about one-third of enrolled participants, minimum 8, maximum 18)

Exclusion Criteria:

* Liver disease other than NAFLD
* Excess alcohol consumption (≥ 2 units/day for women and ≥ 3 units/day for men)
* Current diagnosis of drug induced liver injury
* Receiving drug or placebo in treatment trial now or within 30 days
* Weight loss or gain of ≥ 5 kg in prior 3 months
* Other factors that in the judgment of the principal investigator might preclude study completion
* Women who state they are pregnant. Women who state they are pregnant will be excluded in an abundance of caution, since pregnancy might increase intra-abdominal pressure which in turn might affect the assessment of the different-day reproducibility coefficient of ultrasound and VCTE measurements. Women who state they might be pregnant will be required to do a urine pregnancy test to establish eligibility.
* Patients with active implants such as pacemakers or defibrillators or any other contraindication to ultrasound or VCTE scanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony E Samir, MD, MPH, Principal Investigator — Massachusetts General Hospital; Kathryn Fowler, MD, Principal Investigator — UC San Diego
Locations (2):
- United States (2):
  - UC San Diego, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Pierce TT, Ozturk A, Sherlock SP, Moura Cunha G, Wang X, Li Q, Hunt D, Middleton MS, Martin M, Corey KE, Edenbaum H, Shankar SS, Heymann H, Kamphaus TN, Calle RA, Covarrubias Y, Loomba R, Obuchowski NA, Sanyal AJ, Sirlin CB, Fowler KJ, Samir AE. Reproducibility and Repeatability of US Shear-Wave and Transient Elastography in Nonalcoholic Fatty Liver Disease. Radiology. 2024 Sep;312(3):e233094. doi: 10.1148/radiol.233094. PMID 39254458

RESULTS

PARTICIPANT FLOW:
Groups:
- MGH and UCSD Study Subjects: This study will enroll patients with suspected or confirmed diagnosis of NAFLD. Based on protocol-specified FIB-4 values, about one-third are expected to have low, one-third to have intermediate, and one-third to have high likelihood of advanced fibrosis.
  Sex: 50:50 - Note- no stratification will be done based on sex Age: ≥ 18 yrs Demographic group: Patients with a high probability of NAFLD based on the eligibility criteria General health status: Patients with suspected or confirmed diagnosis of NAFLD Geographic location: Boston, MA (greater metropolitan areas) and San Diego, CA (greater metropolitan areas)
  Ultrasound based shear wave speed and fat quantification methods: Ultrasound based imaging parameters will be collected from all patients in two visits. These will include but may not be limited to SWE results, Quantitative ultrasound parameters,where available,including Attenuation Coefficient, Backscatter Coefficient, Shear Wave Dispersion, Speed of Sound, Ultrasound derived fat fraction Conventional Bmode (gray-scale) and Doppler ultrasound images,including An image of the liver and right kidney on the same image for hepatorenal index calculation Right liver lobe for skin to liver capsule distance calculation Portal vein Doppler for portal vein pulsatility index measurement VCTE and Controlled Attenuation Parameter measurements with the Fibroscan system
Period: Overall Study
Arm/Group | MGH and UCSD Study Subjects
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- MGH and UCSD Study Subjects: NAFLD patients with ultrasound elastography and fat quantification measurements
Arm/Group | MGH and UCSD Study Subjects
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 13
Age, Continuous [Mean (Full Range); unit: years] | 60.4 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Pooled Different-day, Different-operator Reproducibility of Shear Wave Speed Measurements
Description: The same research subject undergoes multiple shear wave elastography measurements (measured in m/s) on multiple ultrasound imaging devices and transient elastography at two visits (baseline + up to 7 days) with different operators. Elastographic measurements are recorded. The median shear wave velocity value (in m/s) is computed for each ultrasound imaging device and is displayed by the transient elastography device. The ultrasound machine measurements are pooled and the pooled different day-different operator reproducibility coefficient for the group of ultrasound machines is computed. The reproducibility coefficient for transient elastography is computed separately. The pooled different-day, different-operator reproducibility coefficient of ultrasound measurements of shear wave speed, is reported in the outcome measure data table section.
Time Frame: (2 visits, baseline + up to 7 days). Outcome measure will be assessed after pooling measurements from all study subjects.
Measure: Number; unit: Reproducibility coefficient (in %)
Units Other Than Participants: SWS measurements on ultrasound images
Groups:
- MGH and UCSD Study Subjects: Ultrasound based shear wave speed (SWS) and transient elastography based SWS measurements were collected from MGH and UCSD study subjects. SWS and transient elastography measurements are obtained in m/s unit.
Arm/Group | MGH and UCSD Study Subjects
Number analyzed (Participants) | 40
Number analyzed (SWS measurements on ultrasound images) | 3600
Reproducibility coefficient (in %) | 30.7

2. Primary Outcome: Different-day, Different-operator Reproducibility Coefficient of Transient Elastography Based Shear Wave Speed Measurements
Description: The same research subject undergoes multiple shear wave elastography measurements (measured in m/s) on multiple ultrasound imaging devices and transient elastography at two visits (baseline + up to 7 days) with different operators. Elastographic measurements are recorded. The median shear wave velocity value (in m/s) is computed for each ultrasound imaging device and is displayed by the transient elastography device. The ultrasound machine measurements are pooled and the pooled different day-different operator reproducibility coefficient for the group of ultrasound machines is computed. The reproducibility coefficient for transient elastography is computed separately. The pooled different-day, different-operator reproducibility coefficient of transient elastography measurements (in m/s unit), is reported in the outcome measure data table section.
Time Frame: (2 visits, baseline + up to 7days). Outcome measure will be assessed after pooling all measurements from all study subjects.
Measure: Number; unit: Reproducibility coefficient (in %)
Units Other Than Participants: SWS measurements on ultrasound images
Groups:
- MGH and UCSD Study Subjects: Transient elastography based SWS measurements were collected from MGH and UCSD study subjects. Transient elastography measurements are obtained in m/s unit.
Arm/Group | MGH and UCSD Study Subjects
Number analyzed (Participants) | 39
Number analyzed (SWS measurements on ultrasound images) | 1170
Reproducibility coefficient (in %) | 35.6

3. Secondary Outcome: Evaluation of Pooled Same-day, Same-operator Repeatability of Shear Wave Speed (SWS)
Description: The same research subject undergoes multiple SWE measurements (in m/s) on multiple devices and transient elastography (TE) at two visits (in 7 days) with different operators. For this outcome measure, the same-day same-operator repeatability is estimated on repeated measurements performed on the same device by the same operator at the same visit. For example, the following structure is followed for a subject; Day1 (Device A, Device B, Device C, TE, Repeated Device A, Repeated Device B), Day2 (Device A, Device B, Device C, TE, Repeated Device C, Repeated TE). The median SWS value (in m/s) is computed for each ultrasound device and is displayed by the TE device. The pooled same-day, same-operator repeatability coefficient of ultrasound measurements of SWS, is reported in the outcome measure data table section.
Time Frame: (2 visits, baseline + up to 7days). Outcome measure will be assessed after pooling measurements from all study subjects.
Measure: Number; unit: Repeatability coefficient (in %)
Units Other Than Participants: SWS measurements on ultrasound images
Arm/Group | MGH and UCSD Study Subjects
Number analyzed (Participants) | 40
Number analyzed (SWS measurements on ultrasound images) | 3600
Repeatability coefficient (in %) | 21

4. Secondary Outcome: Evaluation of Pooled Different-scanner, Same-day Reproducibility of Shear Wave Elastography.
Description: The same research subject undergoes multiple shear wave elastography measurements (measured in m/s) on multiple ultrasound imaging devices and transient elastography at two visits (baseline + up to 7 days) with different operators. The median shear wave velocity value (in m/s) is computed for each ultrasound imaging device and is displayed by the transient elastography device. The reproducibility coefficient of measurements obtained across different ultrasound devices on the same day by the same operator is computed. For example, the following structure is followed for a study subject; Day1 (Device A, Device B, Device C, Transient elastography, Repeated Device A, Repeated Device B), Day2 (Device A, Device B, Device C, Transient elastography, Repeated Device C, Repeated transient elastography).The pooled different-scanner, same-day reproducibility coefficient of ultrasound measurements of SWS, is reported in the outcome measure data table section.
Time Frame: as for outcome 2
Measure: Number; unit: Reproducibility coefficient (in %)
Units Other Than Participants: SWS measurements on ultrasound images
Arm/Group | MGH and UCSD Study Subjects
Number analyzed (Participants) | 40
Number analyzed (SWS measurements on ultrasound images) | 3600
Reproducibility coefficient (in %) | 52.7

5. Secondary Outcome: Evaluation of Same-day, Same-operator Repeatability of Transient Elastography
Description: Same day same operator repeat median TE measures expressed in m/s are compared and the repeatability is estimated. For example, the following structure is followed for a study subject; Day1 (Device A, Device B, Device C, Transient elastography, Repeated Device A, Repeated Device B), Day2 (Device A, Device B, Device C, Transient elastography, Repeated Device C, Repeated transient elastography), which allows estimation of same-day same operator repeatability.
Time Frame: as for outcome 2
Measure: Number; unit: Repeatability coefficient (in %)
Units Other Than Participants: SWS measurements on ultrasound images
Arm/Group | MGH and UCSD Study Subjects
Number analyzed (Participants) | 39
Number analyzed (SWS measurements on ultrasound images) | 1170
Repeatability coefficient (in %) | 19.6

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | MGH and UCSD Study Subjects
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT04828551/Prot_SAP_000.pdf